CLINICAL TRIAL: NCT01258725
Title: Alterations of the Uteroplacental and Fetal Pulmonary Circulation in Patients With Severe Idiopathic Oligohydramnios Following Amnioinfusion Therapy in a Longitudinal Study
Brief Title: Alterations of the Uteroplacental and Fetal Pulmonary Circulation Following Amnioinfusion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Szeged University (Other)
Responsible Party: Attila Pál, University of Szeged, Faculty of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Amnioinfusioncirculation
Record Dates: First submitted 2010-12-07; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Severe Oligohydramnios
Keywords: amnioinfusion, severe idiopahic oligohydramnios
MeSH Terms: conditions — Oligohydramnios

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- amnioinfusion (Experimental): The investigators propose an open trial comparing baseline Doppler waveforms in the uteroplacental and fetal pulmonary circulation in patients presenting with severe, idiopathic olighydramnios (AFI<5, no apparent ethiopathology), managed either with single or with serial amnioinfusions. The patients will be followed up weekly in the fetomaternal unit, Dept. of ObGyn for measuring AFI repeatedly to assess the need for further infusions. These will be carried out when the AFI falls below 5cm again
  Interventions: Procedure: amnioinfusion procedure

INTERVENTIONS:
Procedure: amnioinfusion procedure — Single/serial amnioinfusions aimed at restoring amniotic fluid volume until a normal amount (AFI≥8cm).(Every pregnant women presenting with severe (AFI<5) idiopathic (with unknown origin) oligohydramnios is treated with amnioinfusion at our Dept.)
  Other Names: restoring amniotic fluid volume with intraamniotic transfusion of saline infusion

SUMMARY:
The aim of this study is to compare the uteroplacental and pulmonary circulation of the fetuses with severe (AFI<5cm) idiopathic oligohydramnios (with unknown origin) to those in normal controls. Further purpose of the study is to measure the changes of the uteroplacental and fetal pulmonary circulation in patients presenting with severe idiopathic oligohydramnios, managed either with single amnioinfusion or with serial amnioinfusions.

DETAILED DESCRIPTION:
Severe oligohydramnios (AFI<5) is an uncommon complication of pregnancy and it is often associated with Preterm Premature Rupture of the Membranes (pPROM) or with the lethal congenital abnormality. However, in very few cases it is idiopathic (with no obvious etiopathology) and in the prevention of fetal complication (e.g. pulmonary hypoplasia) the amnioinfusion is a treatment option for the persisting oligohydramnios.

Severe oligohydramnios for >14 days had a predicted mortality rate >90%. Although severe oligohydramnios and pPROM may lead to pulmonary hypoplasia, all of these three factors are independent predictors of pulmonary hypertension. It is obvious that there are some alterations in the fetal pulmonary circulation in cases of severe oligohydramnios.

The preliminary study shows that single/serial amnioinfusion has some beneficial effects on the outcome of the pregnancies complicated with severe idiopathic oligohydramnios: to prolong the gestation, to reduce the number of premature labor and to prevent the adverse neonatal outcome.

The investigators propose an open trial comparing baseline Doppler waveforms in the uteroplacental and fetal pulmonary circulation in patients presenting with severe, idiopathic olighydramnios (AFI<5, no apparent ethiopathology), managed either with single or with serial amnioinfusions and in matched controls (matched in gestational age, parity and gravidity, AFI>8). The patients will be followed up weekly in the fetomaternal unit, Dept. of ObGyn for measuring AFI repeatedly to assess the need for further infusions. These will be carried out when the AFI falls below 5cm again.

Inclusion criteria: Single pregnancy, severe (AFI<4 cm), idiopathic oligohydramnios between the 18 and 34 weeks of gestation. The study is open and will be run by a single ultrasonographer to avoid interobserver bias, and with a set of minimal number of outcome measures recorded. Primary outcome: Doppler waveforms of the uteroplacental and fetal pulmonary circulation.

Alterations in Doppler indices of the Ductus venosus, arteria umbilicalis, arteria uterina, left and right arterial pulmonary branches: (1) systolic/diastolic ratio (S/D), (2) peak systolic velocity; (3) time-averaged velocity; (4) maximum forward velocity during atrial contraction; (5) pulsatility index (PI); (6) Pourcelot's resistance index (RI).

The pulsed Doppler measurements of the arterial pulmonary branches will be carried out from a transverse cross-section of the fetal chest at the level of the cardiac 4-chamber view after visualization with color Doppler. Depending on fetal position, the right or left lung will be examined. Doppler waveforms (sample volume: 0.1-0.3 cm) will be first obtained from the most proximal branch of the pulmonary artery, then in the middle lung region at equal distance from the outer border of the heart and the inner thoracic wall and subsequently in the distal lung region as close as possible to the fetal inner thoracic wall.

Secondary outcomes: Alterations of the Doppler waveforms during the progress of the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years, who are able to consent;
2. Singleton pregnancy;
3. Normal structural examination between 16 and 20 weeks of gestation;
4. Gestation between 18 and 34 weeks (the pregnancy duration determined by ultrasound verification within the 20th week);
5. At least two US examinations at the presentation for confirmation and for the diagnosis of persistent oligohydramnios;
6. Follow up ultrasound examinations weekly in both groups.

Exclusion Criteria:

1. pPROM; 2. Fetal structural anomaly detected at prenatal ultrasonography, or fetal chromosomal abnormalities involving autosomes; 3. Symptoms referring incomplete abortion before 24 weeks of gestation; 4. Maternal contraindications to intervention or prolongation of pregnancy, including severe medical conditions in pregnancy that make the intervention riskful; 5. No active premature labor (shortened cervix <15 mm, <3 cm of cervical dilatation; >6/hour uterine contractions) after 24 weeks of gestation; 6. Cervical cerclage in place; 7. Clear signs of maternal or fetal infection (2 or more of the following: maternal tachycardia >100/min, maternal temperature >38°C, maternal white blood count cells (WBC) >15,000/ml, maternal C-reactive protein (CRP) >20 mg/l, uterine tenderness, foul-smelling vaginal discharge, fetal tachycardia >160 bpm); 8. Suspicion of placental abruption (uterine tenderness and bleeding episodes); 9. Previous invasive procedure in the pregnancy; 10. Fetal condition mandating immediate delivery; 11. Severe bleeding at present; 12. Maternal HIV and HBV/HCV infection; 13. Multiple gestation.

-

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Doppler waveforms of the uteroplacental and fetal pulmonary circulation following amnioinfusion | reaching 34 weeks of gestation

SECONDARY OUTCOMES:
Alterations of the Doppler waveforms during the progress of the pregnancy following amnioinfusion | reaching 34 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: János Sikovanyecz, M.D., Ph.D., Principal Investigator — University of Szeged, Department of Obstetrics and Gynecology; Zoltan Kozinszky, M.D., Ph.D., Study Director — Department of Obstetrics and Gynecology, University of Szeged
Locations (1):
- University of Szeged, Department of Obstetrics and Gynecology, Szeged, Hungary